CLINICAL TRIAL: NCT02394054
Title: Vasopressin's Effect on Behavior and Neural Activity During Social Cognition Tasks
Brief Title: Vasopressin and the Social Brain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Matthew Lieberman, Matthew D. Lieberman, PhD, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 11-003565-3
Record Dates: First submitted 2015-01-22; First posted 2015-03-20 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Social Psychology
Keywords: vasopressin; intranasal administration; healthy sample
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal vasopressin (Experimental): Participants will self-administer 20 IU vasopressin (American Regent Pharmaceuticals). 5 puffs per nostril (1 puff = 2 IU vasopressin).
  Interventions: Drug: Intranasal vasopressin
- Intranasal placebo (Placebo Comparator): 2 mls Glycerine and 3 mls purified water (methylparaben and propylparaben mixed according to purified water formula) for a total of 5 ml, which will be filtered with a 5mu filter. Participants will self-administer 5 puffs per nostril.
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal vasopressin — Through the use of 1oz bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 20 IU vasopressin (American Regent Pharmaceuticals). 5 puffs per nostril (1 puff = 2 IU vasopressin).
  Arms: Intranasal vasopressin
Drug: Intranasal placebo — Through the use of 1oz bottles attached with metered nasal pumps (1 puff = .1ml), participants will self-administer 5 puffs per nostril. Placebo consists of: 2 mls Glycerine and 3 mls purified water (methylparaben and propylparaben mixed according to purified water formula) for a total of 5 ml, which will be filtered with a 5mu filter.
  Arms: Intranasal placebo

SUMMARY:
It has long been established that interpersonal relationships can have a profound impact on health and well-being. Yet, the investigators are still learning about the complex biological processes that contribute to positive social interactions and the ability to develop and maintain social relationships. Recent research has begun to focus on vasopressin, a neuropeptide that is naturally produced in the hypothalamus, because administration of this neuropeptide has been associated with empathy, cooperation, memory of social stimuli (e.g., faces), and brain activity in neural regions associated with social and emotional processes. To date, several aspects of vasopressin's effects on social behavior have been unexplored. As such, the overarching goal of this project is to examine the effects of intranasal vasopressin on several tasks involving learning and social processes. In addition, the investigators will explore associated neural activity through functional magnetic resonance imaging (fMRI). Results from the study will inform our understanding of the neurobiology of socioemotional processes.

The investigators hypothesize that compared to placebo, vasopressin will improve deception detection, increase empathy and altruism, enhance responses to photo stimuli of primary caregivers, and improve learning when the subject has a prosocial goal of teaching another person. These effects will manifest in behavioral and neural activity. It is also hypothesized that main effects will not be found for vasopressin, but rather, analyses of relevant moderators will elucidate these findings.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* Healthy (see below)
* Fluent in English
* Right-handed

Exclusion Criteria:

* Women who gave birth in the last six months, are currently pregnant, planning to become pregnant in the next 6 months, or currently breastfeeding women
* Symptoms of runny nose due to allergies/cold or other reason
* Current restricted fluid intake for any reason
* Heart disease
* Hypertension
* History of myocardial infarction
* History of cardiac arrhythmia
* Kidney or liver disease
* Vascular disease
* Epilepsy
* Migraine
* Asthma
* Nephritis
* Diabetes and other endocrine diseases
* Frequent or unexplained fainting
* History of stroke
* Aneurysm or brain hemorrhage
* Active psychiatric diagnosis
* Current psychopharmacologic treatment
* Drug or alcohol abuse
* Medical or neurological illness
* Regular use of medication (e.g., vasoconstrictive medications)
* Medication intake less than 2 weeks prior to study (5 weeks for fluoxetine) including daily non-steroidal anti-inflammatory drugs
* Smoking more than 15 cigarettes a day
* Consumption of any alcoholic beverages in the past 24 hours will be excluded
* Elevated blood pressure (>135/90)
* Low blood pressure (<90/55)
* Body temperature >100.1 F
* Left-handed
* Claustrophobia
* Presence of metal in their body

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Changes in neural brain activity, as observed by fMRI, when observing others during social inclusion vs. exclusion | Between 40-115 minutes post administration
  Whole brain and region of interest (ROI) regression analysis will be used to compare the neural activity of participants in the vasopressin/placebo groups. A design matrix will be created for each participant, modeling activity that is greater during the exclusion portion of the cyberball task (Williams et al., 2012) versus the inclusion portion. A first-level analysis will compare [(friend exclusion>friend inclusion)>(stranger exclusion>stranger inclusion)] for each participant. A second-level group analysis will compare these first-level contrasts between the vasopressin and placebo groups.

SECONDARY OUTCOMES:
Ratings of empathic concern after witnessing social exclusion in a friend or a stranger | Between 40-115 minutes post administration
  Ratings of empathic concern will be calculated for each participant by deriving a composite from self-report ratings of sympathy and compassion. Using a mixed 2 (friend, stranger) x 2 (vasopressin, placebo) factorial design, comparisons of these ratings will then be made for those in the vasopressin vs. placebo groups. Main effects of drug condition (vasopressin, placebo) as well as the interaction between drug condition and target (friend, stranger) will be analyzed at a significance level of p<.05.
Altruism and punishment as measured by number of points given to excluders and those excluded | Between 40-115 minutes post administration
  Ratings of altruism and punishment will be calculated by examining how many point (1-10) participants decide to allocate towards the friend-excluder, stranger-excluder, excluded friend, and excluded stranger after watching each social exclusion game. Using a mixed 2 (friend, stranger) x 2 (vasopressin, placebo) factorial design, comparisons of these ratings will then be made for those in the vasopressin vs. placebo groups. Main effects of drug condition (vasopressin, placebo) and target (friend, stranger), as well as an interaction between drug condition and target will be analyzed at a significance level of p<.05.
Changes in neural brain activity, as observed by fMRI, while attempting to detect deception | Between 40-115 minutes post administration
  Whole brain and region of interest (ROI) regression analysis will be used to compare the neural activity of participants in the vasopressin/placebo groups. A design matrix will be created for each participant, modeling activity that is greater during the deception detection task versus a control task. A first-level analysis will compare deception-detection>control for each participant. A second-level group analysis will compare this first-level contrast between the vasopressin and placebo groups.
Accuracy of deception detection as measured by self-report | Between 40-115 minutes post administration
  The investigators will compare the percentage of correct deception detection trials for participants in the vasopressin group to those in the placebo group by running a two-tailed t-test with a statistical cutoff of p<.05 to determine significance.
Changes in neural brain activity, as observed by fMRI, when viewing images of primary caregivers versus strangers | Between 40-115 minutes post administration
  Whole brain and region of interest (ROI) regression analysis will be used to compare the neural activity of participants in the vasopressin/placebo groups. A design matrix will be created for each participant, modeling activity that is greater while viewing photo stimuli of ones primary caregivers versus viewing photo stimuli of matched strangers. A first-level analysis will compare primary-caregiver-viewing>stranger-viewing for each participant. A second-level group analysis will compare this first-level contrast between the vasopressin and placebo groups.
Changes in brain neural activity, observed by fMRI, in response to a reading comprehension task | Between 40-90 minutes post administration
  Whole brain and region of interest (ROI) regression analysis will be used to compare the neural activity of participants in the tutor/memorizer and vasopressin/placebo groups. A design matrix will be created for each participant, modeling activity that is greater during reading comprehension compared with the grammar control passage. First level analyses will compare the response during the reading comprehension passages relative to the grammar control passages. Second level group analyses will compare the first level contrasts between the tutor vs. memorizer groups as well as the vasopressin vs. placebo groups. In regression analyses the investigators will enter each participant's comprehension test score in the tutor and then memorizer condition as a regressor in a whole-brain and ROI analysis to determine which brain regions were more active during the encoding of the reading comprehension passage compared to the grammar control passage.
Performance on a memory test of reading comprehension as measured by percentage of questions answered correctly | Between 40-90 minutes post administration
  Accuracy will be calculated for each participant by dividing the number of correct responses by the total number of questions. The investigators will then conduct a between-subjects 2x2 ANOVA on the accuracy scores for the four groups of interest (i.e., vasopressin-tutor, vasopressin-memorizer, placebo-tutor, placebo-memorizer). A significance level of p<.05 will be used to determine whether there are significant differences between the groups. The investigators will examine whether there is a main effect of either factor (vasopressin vs. placebo, tutor vs. memorize) as well as an interaction between the factors of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Lieberman, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Department of Psychology, Los Angeles, California, United States

REFERENCES:
- [Derived] Straccia MA, Teed AR, Katzman PL, Tan KM, Parrish MH, Irwin MR, Eisenberger NI, Lieberman MD, Tabak BA. Null results of oxytocin and vasopressin administration on mentalizing in a large fMRI sample: evidence from a randomized controlled trial. Psychol Med. 2023 Apr;53(6):2285-2295. doi: 10.1017/S0033291721004104. Epub 2021 Oct 15. PMID 37310308